CLINICAL TRIAL: NCT03342781
Title: Using a High-flow Nasal Cannula Provided Superior Results to Diffuser Delivery in Severe Bronchiolitis: a Prospective, Randomized Controlled Study
Brief Title: Using HFNC in Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Betul Ergul, Principal Investigator, Kayseri Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/504
Record Dates: First submitted 2017-11-02; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Respiratory Failure; Bronchiolitis
Keywords: bronchiolitis; diffuser mask; high-flow nasal oxygen; pediatric intensive-care unit
MeSH Terms: conditions — Respiratory Insufficiency; Bronchiolitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diffuser-mask group (Active Comparator): The patients received oxygen therapy (8-15 L/min) from an OxyMask (Southmedic, Inc., Barrie, ON, Canada) to maintain oxygen saturation (SpO2) > 92%. Oxygen therapy was halted if SpO2 was maintained at a level greater than 92% for more than 4 h. The oxygen flow rate was then decreased to 2 L/min and the patient was monitored while breathing room air.
  Interventions: Device: Diffuser oxygen mask
- HFNC group (Active Comparator): The patients received oxygen therapy at a high flow rate from a Precision Flow nasal cannula (Vapotherm, Inc., Stevensville, MD, USA). We selected a 1.9 mm pediatric cannula, which can dispense 1-20 L/min of oxygen. The initial oxygen flow rate was 1 L/kg/min and the FiO2 was 100%. The initial flow rate was increased by 1 L/kg/min until the SpO2 reached 92%. The initial FiO2 was decreased once the SpO2 was greater than 92% and the oxygen flow rate was maintained. HFNC therapy was halted if SpO2 was maintained at a level greater than 92% for more than 4 h at a FiO2 value of 21%, and the patient was transferred to a ward.
  Interventions: Device: high flow nasal oxygen therapy

INTERVENTIONS:
Device: high flow nasal oxygen therapy — Oxygen therapy using a high-flow nasal cannula (HFNC) is a high-flow oxygen delivery system that enhances the efficiency of respiration by using high flow rates to clear dead space and provide fresh oxygen. This system supplies oxygen at a high flow rate through a loose nasal cannula.
  Arms: HFNC group
Device: Diffuser oxygen mask — diffuser mask is a low-flow delivery system, which is capable of delivering up to 90% of the fraction of inspired oxygen (FiO2) with low CO2 retention. In this system, the FiO2 can be adjusted by modifying the flow velocity to deliver the quantity of oxygen that the patient requires. Oxygen is supplied to the patient in a jet that flows from a device mounted on the oxygen mask. This ensures that a high concentration of oxygen is provided at a low flow rate.
  Arms: Diffuser-mask group

SUMMARY:
The investigators compared oxygen therapy using the HFNC and diffuser mask (an effective low-flow oxygen delivery system) to treat patients with moderate-to-severe acute bronchiolitis admitted to an intensive care unit (ICU).

DETAILED DESCRIPTION:
Acute bronchiolitis results from inflammation of the bronchioles and is usually caused by a viral infection. It is most common in children younger than 2 years old and is one of the most frequent reasons why a child is admitted to hospital. There is no established, specific therapy for acute bronchiolitis and it is commonly treated using supplemental oxygen and by ensuring that the patient remains hydrated.

Oxygen therapy can be applied using a low- or high-flow oxygen delivery system. For example, a diffuser mask (OxyMask) is a low-flow delivery system, which is capable of delivering up to 90% of the fraction of inspired oxygen (FiO2) with low carbon dioxide (CO2) retention. In this system, the FiO2 can be adjusted by modifying the flow velocity to deliver the quantity of oxygen that the patient requires. Oxygen is supplied to the patient in a jet that flows from a device mounted on the oxygen mask. This ensures that a high concentration of oxygen is provided at a low flow rate. Additionally, CO2 retention is minimal because the mask has a fenestrated structure. Therefore, a diffuser mask is a more effective oxygen delivery method than many other low-flow delivery systems including the nasal cannula and simple oxygen mask.

Oxygen therapy using a high-flow nasal cannula (HFNC) is a high-flow oxygen delivery system that enhances the efficiency of respiration by using high flow rates to clear dead space and provide fresh oxygen. This system supplies oxygen at a high flow rate through a loose nasal cannula. HFNC therapy provides heated and humidified oxygen to fill the dead space in the nasopharynx and produces minimal positive airway pressure. It enhances the passage of air through the airway by reducing inspiratory pressure. Previous studies have demonstrated that using a HFNC can decrease respiratory effort and improve gas exchange. In recent years, many studies have suggested that high-flow nasal oxygen therapy is more effective than low-flow systems. This is substantiated by significant decreases in the use of mechanical ventilation since HFNC therapy was introduced.

Previous reports on the effectiveness of HFNC therapy in treating acute bronchiolitis have come primarily from observational work and there are few relevant, randomized controlled studies. Additionally, previous studies have compared HFNC therapy with less effective, low-flow systems (e.g., the simple mask or nasal cannula). To the best of our knowledge, no randomized controlled trial has compared the effectiveness of the HFNC and diffuser mask in treating bronchiolitis.

In this study, the investigators compared oxygen therapy using the HFNC and diffuser mask (an effective low-flow oxygen delivery system) to treat patients with moderate-to-severe acute bronchiolitis admitted to an intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Included patients were aged between 1 and 24 months and had been diagnosed with moderate or severe acute bronchiolitis. They were admitted to the ICU, requiring supplemental oxygen, because their SpO2 measurements were less than 94% while breathing room air.

Exclusion Criteria:

* Any patients requiring immediate respiratory support (non-invasive or invasive mechanical ventilation, altered mental status, or apnea at presentation), those already admitted to the ICU due to respiratory failure, those with underlying chronic lung disease or cardiovascular disorders, those with obstructions of the upper respiratory tract, and those with cranial malformations were excluded.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-03-01; Primary Completion 2016-12-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
presence of treatment failure | up to 1 month
  Treatment failure was defined as meeting two of the following criteria [16]:
  1. No change or an increase in respiration rate compared with baseline.
  2. No change or an increase in heart rate compared with baseline.
  3. Persistence of low SpO2 (<%92) measurements despite an adequate oxygen flow rate and FiO2 in the HFNC group/oxygen flow rate of 15 L/min in the mask group.

SECONDARY OUTCOMES:
total duration of oxygen therapy | up to 1 month
Length of hospital stay day | up to 1 month
time of treatment failure | up to 1 month

REFERENCES:
- [Background] Tapiainen T, Aittoniemi J, Immonen J, Jylkka H, Meinander T, Nuolivirta K, Peltola V, Salo E, Seuri R, Walle SM, Korppi M. Finnish guidelines for the treatment of laryngitis, wheezing bronchitis and bronchiolitis in children. Acta Paediatr. 2016 Jan;105(1):44-9. doi: 10.1111/apa.13162. Epub 2015 Nov 6. PMID 26295564
- [Background] Kose S, Sehriyaroglu A, Esen F, Ozdemir A, Kardas Z, Altug U, Karakus E, Ozcan A, Kisaarslan AF, Elmali F, Torun YA, Kose M. Comparing the Efficacy of 7%, 3% and 0.9% Saline in Moderate to Severe Bronchiolitis in Infants. Balkan Med J. 2016 Mar;33(2):193-7. doi: 10.5152/balkanmedj.2016.16840. Epub 2016 Mar 1. PMID 27403389
- [Background] Paul JE, Hangan H, Hajgato J. The OxyMask() development and performance in healthy volunteers. Med Devices (Auckl). 2009;2:9-17. Epub 2008 Dec 11. PMID 22915909
- [Background] Beecroft JM, Hanly PJ. Comparison of the OxyMask and Venturi mask in the delivery of supplemental oxygen: pilot study in oxygen-dependent patients. Can Respir J. 2006 Jul-Aug;13(5):247-52. doi: 10.1155/2006/720320. PMID 16896425
- [Background] Ling E, McDonald L, Dinesen TR, DuVall D. The OxyArm - a new minimal contact oxygen delivery system for mouth or nose breathing. Can J Anaesth. 2002 Mar;49(3):297-301. doi: 10.1007/BF03020531. PMID 11861350
- [Background] Bressan S, Balzani M, Krauss B, Pettenazzo A, Zanconato S, Baraldi E. High-flow nasal cannula oxygen for bronchiolitis in a pediatric ward: a pilot study. Eur J Pediatr. 2013 Dec;172(12):1649-56. doi: 10.1007/s00431-013-2094-4. Epub 2013 Jul 31. PMID 23900520
- [Background] Pham TM, O'Malley L, Mayfield S, Martin S, Schibler A. The effect of high flow nasal cannula therapy on the work of breathing in infants with bronchiolitis. Pediatr Pulmonol. 2015 Jul;50(7):713-20. doi: 10.1002/ppul.23060. Epub 2014 May 21. PMID 24846750
- [Background] Hough JL, Pham TM, Schibler A. Physiologic effect of high-flow nasal cannula in infants with bronchiolitis. Pediatr Crit Care Med. 2014 Jun;15(5):e214-9. doi: 10.1097/PCC.0000000000000112. PMID 24705569
- [Background] Keenan SP, Sinuff T, Cook DJ, Hill NS. Does noninvasive positive pressure ventilation improve outcome in acute hypoxemic respiratory failure? A systematic review. Crit Care Med. 2004 Dec;32(12):2516-23. doi: 10.1097/01.ccm.0000148011.51681.e2. PMID 15599160
- [Background] ten Brink F, Duke T, Evans J. High-flow nasal prong oxygen therapy or nasopharyngeal continuous positive airway pressure for children with moderate-to-severe respiratory distress?*. Pediatr Crit Care Med. 2013 Sep;14(7):e326-31. doi: 10.1097/PCC.0b013e31828a894d. PMID 23842586
- [Background] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312